CLINICAL TRIAL: NCT03898752
Title: Is Oxidative Stress in Semen Reduced by Lifestyle Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Humaidan (Other)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, MD, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MiOxysis_Skive
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Oligospermia
MeSH Terms: conditions — Oligospermia | interventions — Docosahexaenoic Acids; coenzyme Q10; Geritol

STUDY DESIGN:
Intervention Model Description: All men with DFI >15 (SCSA method) are assigned to life-style intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle intervention (Experimental): Diet, omega-3 fish oil (1g daily), CoQ10 (100 mg/day) and a normal Multi-vitamin, Smoking cessation, weight loss, exercise,
  Interventions: Dietary Supplement: Omega 3

INTERVENTIONS:
Dietary Supplement: Omega 3 — Omega 3: 1g daily for 3 months CoQ10: 100 mg daily for 3 months Multivitamin: 1 normal multivitamin tablet daily for 3 months
  Other Names: Coenzyme Q10 (CoQ10); Multi-vitamin

SUMMARY:
In this study we aim to investigate whether a 3-month life-style intervention would reduce oxidative stress (OS) in semen in men of infertile couples attending IVF-treatment. Men with a DFI above 15% (SCSA method) are recruited for intervention with a 3-month follow-up.

It is hypothesized that men who also have a OS above 1.34 using a novel OS diagnostic method (MiOXSYS) respond better to antioxidant treatment with a change in OS and DFI. The primary outcome is the change in OS following the intervention. Secondary outcomes are morphological semen parameters and DNA fragmentation index.

ELIGIBILITY:
Inclusion Criteria:

* DFI>15
* Attending IVF treatment for unknown or male factor infertility.

Exclusion Criteria:

* Genetic diseases
* Azospermia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Oxidative stress | 3 months
  Oxidative stress as measured with MiOxysis (Ayto Bioscience inc).

SECONDARY OUTCOMES:
Semen quality | 3 months
  Morphological semen parameters using WHO recommendation for semen analysis.
DNA fragmentation index | 3 months
  DNA fragmentation index as measured by the method by SPZlab A/S (SCSA method)

CONTACTS AND LOCATIONS:
Locations (1):
- The Fertility Clinic Skive, Skive, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Not allowed by Danish legislation to publish individual meta-data.

REFERENCES:
- [Derived] Humaidan P, Haahr T, Povlsen BB, Kofod L, Laursen RJ, Alsbjerg B, Elbaek HO, Esteves SC. The combined effect of lifestyle intervention and antioxidant therapy on sperm DNA fragmentation and seminal oxidative stress in IVF patients: a pilot study. Int Braz J Urol. 2022 Jan-Feb;48(1):131-156. doi: 10.1590/S1677-5538.IBJU.2021.0604. PMID 34472769